CLINICAL TRIAL: NCT03077620
Title: Sleep Quality and Amyloid-Beta Kinetics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 201602165
Record Dates: First submitted 2016-10-17; First posted 2017-03-13 (Actual); Results first posted 2022-05-17 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Amyloid-beta
MeSH Terms: conditions — Plaque, Amyloid | interventions — suvorexant; Sugars

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (4):
- Poor sleep group treatment 1 (Experimental): 10mg Suvorexant tablet h.s. for two consecutive nights
  Interventions: Drug: Suvorexant
- Poor sleep group control (Placebo Comparator): Participant will receive placebo for two consecutive nights and sleep as normal under the same controlled conditions in a clinical research unit.
  Interventions: Drug: Placebo
- Good sleep group (Placebo Comparator): Participant will receive placebo for two consecutive nights and sleep as normal under the same controlled conditions in a clinical research unit.
  Interventions: Drug: Placebo
- Poor sleep group treatment 2 (Experimental): 20mg Suvorexant tablet h.s. for two consecutive nights
  Interventions: Drug: Suvorexant

INTERVENTIONS:
Drug: Suvorexant — Participants will be given a sleep aid (10mg or 20mg suvorexant) at bedtime for two consecutive nights that they are spending in a research unit.
  Other Names: Belsomra
  Arms: Poor sleep group treatment 1; Poor sleep group treatment 2
Drug: Placebo — Participants will be given a placebo at bedtime for two consecutive nights that they are spending in a research unit.
  Other Names: sugar pill
  Arms: Good sleep group; Poor sleep group control

SUMMARY:
The purpose of this study is to change the concentration of amyloid-beta in human cerebrospinal fluid (CSF) by modification of sleep efficiency.

DETAILED DESCRIPTION:
The purpose of the study is to investigate whether or not increasing sleep efficiency will change the concentration of amyloid-beta in cerebrospinal fluid (CSF).

ELIGIBILITY:
Inclusion Criteria:

* Age 45-65 years
* Any sex
* Any race/ethnicity
* Mini-Mental Status Examination score (MMSE) >=27
* Sleep efficiency measured by actigraphy to determine good sleeper or poor sleeper

Exclusion Criteria:

* Cognitive impairment as determined by history of MMSE < 27
* Inability to speak or understand English
* BMI >35
* Any sleep disorders other than insomnia
* history of sleep-disordered breathing
* STOP-Bang score > 3
* History or reported symptoms suggestive of restless legs syndrome, narcolepsy or other sleep disorders
* Sleep schedule outside the range of bedtime 8PM-12AM and wake time 4AM-9AM
* Contraindication to lumbar catheter (anticoagulants; bleeding disorder; allergy to lidocaine or disinfectant; prior central nervous system or lower back surgery)
* Cardiovascular disease requiring medication except for controlled hypertension (PI discretion)
* Stroke
* Hepatic or renal impairment
* Pulmonary disease (PI discretion)
* Type 1 diabetes
* HIV or AIDS
* Neurologic or psychiatric disorder requiring medication (PI discretion)
* Alcohol or tobacco use (PI discretion)
* Use of sedating medications
* Inability to get out of bed independently
* Abnormal movement of the non-dominant arm (would affect actigraphy data in unpredictable ways)
* Abnormal physical examination
* Current pregnancy
* History of migraine headaches (PI discretion)
* History of drug abuse in the past 6 months
* Urinary or fecal incontinence
* Difficulty sleeping in an unfamiliar environment (good sleep quality group only)
* History or presence of any clinically significant medication condition, behavioral or psychiatric condition (including suicidal ideation), or surgical history based on medical record or patient report that could affect the safety of the subject or interfere with study assessments or in the judgment of the PI is not a good candidate

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2021-03-28 (Actual); Study Completion 2021-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Lucey, MD, Principal Investigator — Washington University Medical School
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Poor Sleep Group Control | Poor Sleep Group Treatment 1 | Poor Sleep Group Treatment 2 | Good Sleep Group
Started | 14 | 14 | 14 | 6
Completed | 13 | 13 | 12 | 6
Not Completed | 1 | 1 | 2 | 0
Not completed — Unable to place lumbar catheter | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: There was a 6th participant in the Good sleep group that had a lumbar catheter placed. However, minimal CSF was collected at a majority of the timepoints. There was insufficient samples of CSF collected to measure amyloid-beta (minimum volume needed was 0.5 ml at each timepoint). The participant agreed to continue the study for collection of blood and to try and continue collecting CSF, but would not agree to replacing the lumbar catheter.
Groups:
- Total: Total of all reporting groups
Arm/Group | Poor Sleep Group Control | Poor Sleep Group Treatment 1 | Poor Sleep Group Treatment 2 | Good Sleep Group | Total
Number analyzed (Participants) | 13 | 13 | 12 | 5 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 12 | 5 | 43
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.94 (6.1) | 56.95 (4.35) | 54.30 (5.66) | 59.18 (7.24) | 56.23 (5.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 9 | 5 | 31
  Male | 5 | 4 | 3 | 0 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 1 | 0 | 8
  White | 10 | 9 | 11 | 5 | 35
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 13 | 12 | 5 | 43

OUTCOME MEASURES:

1. Primary Outcome: Difference in Amyloid-beta (Abeta) Concentration in the CSF (Cerebral Spinal Fluid) of Individuals With Poor Sleep Efficiency Compared to Those With Good Sleep Efficiency as Measured by ng/ml
Description: Mean difference in amyloid-beta-42 concentration between individuals with poor sleep efficiency (Poor sleep group control) compared to those with good sleep efficiency (Good sleep group)
Time Frame: 36 hours of CSF collection
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Poor Sleep Group Control | Good Sleep Group
Number analyzed (Participants) | 13 | 5
ng/ml
  Amyloid-beta-42 concentration at hour 0 (ng/ml) | 0.573 (0.206) | 0.623 (0.189)
  Amyloid-beta-42 concentration at hour 2 (ng/ml) | 0.600 (0.232) | 0.520 (0.168)
  Amyloid-beta-42 concentration at hour 4 (ng/ml) | 0.583 (0.180) | 0.528 (0.171)
  Amyloid-beta-42 concentration at hour 6 (ng/ml) | 0.573 (0.155) | 0.542 (0.174)
  Amyloid-beta-42 concentration at hour 8 (ng/ml) | 0.598 (0.189) | 0.548 (0.155)
  Amyloid-beta-42 concentration at hour 10 (ng/ml) | 0.602 (0.173) | 0.537 (0.149)
  Amyloid-beta-42 concentration at hour 12 (ng/ml) | 0.635 (0.205) | 0.536 (0.129)
  Amyloid-beta-42 concentration at hour 14 (ng/ml) | 0.645 (0.203) | 0.556 (0.126)
  Amyloid-beta-42 concentration at hour 16 (ng/ml) | 0.661 (0.196) | 0.578 (0.139)
  Amyloid-beta-42 concentration at hour 18 (ng/ml) | 0.659 (0.184) | 0.579 (0.131)
  Amyloid-beta-42 concentration at hour 20 (ng/ml) | 0.680 (0.195) | 0.568 (0.123)
  Amyloid-beta-42 concentration at hour 22 (ng/ml) | 0.674 (0.203) | 0.584 (0.137)
  Amyloid-beta-42 concentration at hour 24 (ng/ml) | 0.691 (0.177) | 0.618 (0.148)
  Amyloid-beta-42 concentration at hour 26 (ng/ml) | 0.674 (0.198) | 0.592 (0.123)
  Amyloid-beta-42 concentration at hour 28 (ng/ml) | 0.692 (0.191) | 0.658 (0.155)
  Amyloid-beta-42 concentration at hour 30 (ng/ml) | 0.660 (0.183) | 0.680 (0.099)
  Amyloid-beta-42 concentration at hour 32 (ng/ml) | 0.652 (0.194) | 0.621 (0.162)
  Amyloid-beta-42 concentration at hour 34 (ng/ml) | 0.682 (0.201) | 0.620 (0.146)
  Amyloid-beta-42 concentration at hour 36 (ng/ml) | 0.743 (0.183) | 0.625 (0.143)
Statistical Analysis 1: Comparison: Poor Sleep Group Control vs Good Sleep Group; Test type: Superiority; p = 0.05, Mixed Models Analysis — Poor sleepers compared to good sleepers with Compound Symmetry covariance structure. Mean difference is poor sleepers minus good sleepers; Mean Difference (Final Values) = 0.119, 95% CI 2-sided [-0.017 to 0.256], Standard Error of Mean 0.064

2. Primary Outcome: Difference in Amyloid-beta (Abeta) Concentration in the CSF (Cerebral Spinal Fluid) of Individuals With Poor Sleep Efficiency Treated With Placebo, Suvorexant 10 mg, or Suvorexant 20 mg as Measured by ng/ml
Description: Mean difference in amyloid-beta-42 concentration between individuals with poor sleep efficiency who were treated with placebo (Poor sleep group control), Suvorexant 10 mg (Poor sleep group treatment 1), and Suvorexant 20 mg (Poor sleep group treatment 2)
Time Frame: 36 hours of CSF collection
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Poor Sleep Group Control | Poor Sleep Group Treatment 1 | Poor Sleep Group Treatment 2
Number analyzed (Participants) | 13 | 13 | 12
ng/ml
  Amyloid-beta-42 concentration at hour 0 (ng/ml) | 0.573 (0.206) | 0.519 (0.171) | 0.648 (0.146)
  Amyloid-beta-42 concentration at hour 2 (ng/ml) | 0.600 (0.232) | 0.520 (0.182) | 0.648 (0.129)
  Amyloid-beta-42 concentration at hour 4 (ng/ml) | 0.583 (0.180) | 0.536 (0.205) | 0.679 (0.129)
  Amyloid-beta-42 concentration at hour 6 (ng/ml) | 0.573 (0.155) | 0.544 (0.207) | 0.678 (0.139)
  Amyloid-beta-42 concentration at hour 8 (ng/ml) | 0.598 (0.189) | 0.546 (0.217) | 0.670 (0.122)
  Amyloid-beta-42 concentration at hour 10 (ng/ml) | 0.602 (0.173) | 0.544 (0.222) | 0.679 (0.124)
  Amyloid-beta-42 concentration at hour 12 (ng/ml) | 0.635 (0.205) | 0.558 (0.222) | 0.660 (0.121)
  Amyloid-beta-42 concentration at hour 14 (ng/ml) | 0.645 (0.203) | 0.583 (0.223) | 0.679 (0.111)
  Amyloid-beta-42 concentration at hour 16 (ng/ml) | 0.661 (0.196) | 0.619 (0.233) | 0.685 (0.120)
  Amyloid-beta-42 concentration at hour 18 (ng/ml) | 0.659 (0.184) | 0.614 (0.205) | 0.697 (0.140)
  Amyloid-beta-42 concentration at hour 20 (ng/ml) | 0.680 (0.195) | 0.615 (0.197) | 0.707 (0.139)
  Amyloid-beta-42 concentration at hour 22 (ng/ml) | 0.674 (0.203) | 0.631 (0.199) | 0.776 (0.161)
  Amyloid-beta-42 concentration at hour 24 (ng/ml) | 0.691 (0.177) | 0.646 (0.198) | 0.738 (0.158)
  Amyloid-beta-42 concentration at hour 26 (ng/ml) | 0.674 (0.198) | 0.653 (0.193) | 0.737 (0.169)
  Amyloid-beta-42 concentration at hour 28 (ng/ml) | 0.692 (0.191) | 0.652 (0.191) | 0.759 (0.166)
  Amyloid-beta-42 concentration at hour 30 (ng/ml) | 0.660 (0.183) | 0.631 (0.189) | 0.707 (0.125)
  Amyloid-beta-42 concentration at hour 32 (ng/ml) | 0.652 (0.194) | 0.627 (0.215) | 0.726 (0.16)
  Amyloid-beta-42 concentration at hour 34 (ng/ml) | 0.682 (0.201) | 0.627 (0.226) | 0.714 (0.159)
  Amyloid-beta-42 concentration at hour 36 (ng/ml) | 0.743 (0.183) | 0.624 (0.217) | 0.724 (0.126)
Statistical Analysis 1: Comparison: Poor Sleep Group Control vs Poor Sleep Group Treatment 1; Test type: Superiority; p = 0.05, Mixed Models Analysis — After corrected for multiple comparisons with Bonferroni test, treatment groups 1 and 2 compared to placebo with Compound Symmetry covariance structure. Mean difference is placebo minus treatment group; Mean Difference (Final Values) = 0.004, 95% CI 2-sided [-0.078 to 0.087], Standard Error of Mean 0.033
Statistical Analysis 2: Comparison: Poor Sleep Group Control vs Poor Sleep Group Treatment 2; Test type: Superiority; p = 0.05, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 0.033, 95% CI 2-sided [-0.051 to 0.117], Standard Error of Mean 0.033

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from when the participants were consented into the study until 48 hours after the lumbar catheter was removed (~3 months).
Arm/Group | Poor Sleep Group Control | Poor Sleep Group Treatment 1 | Poor Sleep Group Treatment 2 | Good Sleep Group
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13 | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/12 | 0/6
Other Adverse Events (participants affected / at risk) | 10/13 | 10/13 | 10/12 | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Poor Sleep Group Control (N=13) | Poor Sleep Group Treatment 1 (N=13) | Poor Sleep Group Treatment 2 (N=12) | Good Sleep Group (N=6)
Headache (Nervous system disorders) | 10 (10) | 7 (7) | 9 (9) | 2 (2)
Headache requiring blood patch (Nervous system disorders) | 2 (2) | 5 (5) | 2 (2) | 0 (0) — Headache requiring blood patch after removal of lumbar catheter
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0)
Presyncope with lumbar catheter placement (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Back/neck pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6) | 7 (7) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash, swelling, or bruising at lumbar catheter site (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Ringing in ears (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-03): https://cdn.clinicaltrials.gov/large-docs/20/NCT03077620/Prot_SAP_000.pdf